CLINICAL TRIAL: NCT00144300
Title: A Two Year Open Label, Randomized, Parallel Group, Blinded Assessment Ophthalmologic Safety Study of Pramipexole IR Versus Ropinirole in Early Parkinson's Disease Patients
Brief Title: Ophthalmologic Safety Study of Pramipexole Immediate Release (IR) Versus Ropinirole in Early Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 248.538
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; ropinirole

ARMS (2):
- Mirapex (Active Comparator): Mirapex tablets three times daily (TID) dosing according to manufacturer's guidelines
  Interventions: Drug: Mirapex
- Requip (Active Comparator): Requip tablets three times daily (TID) dosing according to manufacturer's guidelines
  Interventions: Drug: Requip

INTERVENTIONS:
Drug: Mirapex — Standard marketed product dispensed according to manufacturer's guidelines
  Arms: Mirapex
Drug: Requip — Standard marketed product dispensed according to manufacturer's guidelines
  Arms: Requip

SUMMARY:
To determine if there is any difference in the presence of retinal deterioration in PD patients treated with pramipexole IR versus ropinirole as monitored by comprehensive ophthalmologic assessments from baseline to the end of study at two years.

ELIGIBILITY:
Inclusion criteria

Diagnosis and main criteria for inclusion. Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Patients with idiopathic Parkinson's disease of less than 7 years characterized as Stage I-III by the Modified Hoehn and Yahr Scale and with a maximum of 6 months cumulative lifetime exposure to levodopa and/or dopamine agonist. Patients on current dopamine agonist therapy would require 14-day washout.
2. Age at least 30 years.
3. Women of childbearing potential must have a negative serum beta-HCG pregnancy test at the Screen (Baseline) visit and the patient must use adequate contraceptive methods.
4. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
5. Patients who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.

Exclusion criteria

Main criteria for exclusion. The presence of any of the following would make a patient ineligible for enrollment into the study:

1. Previous history of allergic response or complications with any dopaminergic agonist drug
2. Atypical PD syndromes
3. History of stereotactic brain surgery
4. Positive hepatitis B (surface antigen) or hepatitis C (antibody)
5. Surgery within 180 days of randomization which would negatively impact participation
6. Folstein's Mini Mental State Examination (MMSE) score of 24 or less
7. History of active epilepsy (seizure) in the past 1 year
8. Third degree AV block or sick sinus syndrome
9. Congestive heart failure, Class III or IV
10. Unstable heart disease such as unstable angina, dysrhythmia, or myocardial infarction in prior 6 months
11. Symptomatic orthostatic hypotension
12. Clinically significant liver disease or renal disease
13. Malignant melanoma or history of previously treated malignant melanoma.
14. Prohibited medications taken (including any drug known to have potential retino-toxic effects taken in the prior 12 months; neuroleptics taken within prior 6 months, MAO inhibitors except rasagiline or selegiline taken within prior 3 months, beta-blockers taken to treat Parkinson's disease in the prior 30 days, and Coenzyme Q10 taken within 14 days)
15. Albinism/Albinoidism of any degree, type or syndrome
16. History of glaucoma with or without treatment
17. Inherited or acquired retinopathy such as age-related macular degeneration with visual loss
18. Sarcoidosis
19. Diabetes mellitus of any degree even if diet or insulin controlled
20. Best corrected visual acuity (BCVA) of less than 20/40 by ETDRS
21. Refractive error of greater than minus-6 diopters
22. Abnormal electroretinogram (ERG)
23. Unable to dilate pupils
24. History of severe eye trauma that might affect the outcome of the study
25. History of psychosis
26. Participation in other investigational drug studies or use of investigational drugs within prior 30 days

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2005-01; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (21):
- United States (21):
  - 248.538.00007 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 248.538.00008 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 248.538.00021 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 248.538.00022 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 248.538.00001 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 248.538.00002 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 248.538.00016 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.538.00023 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 248.538.00013 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 248.538.00009 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 248.538.00011 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.538.00005 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 248.538.00014 Boehringer Ingelheim Investigational Site, Southfield, Michigan
  - 248.538.00010 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.538.00015 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.538.00020 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.538.00012 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 248.538.00006 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 248.538.00004 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 248.538.00003 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.538.00017 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Seiple W, Jennings D, Rosen RB, Borchert L, Canale L, Fagan N, Gordon MF. Ophthalmologic Baseline Characteristics and 2-Year Ophthalmologic Safety Profile of Pramipexole IR Compared with Ropinirole IR in Patients with Early Parkinson's Disease. Parkinsons Dis. 2016;2016:8298503. doi: 10.1155/2016/8298503. Epub 2016 Dec 18. PMID 28078162

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: Flexible: 0.125 mg 3 times daily up to maximum tolerated
- Ropinirole: Flexible: 0.25 mg 3 times daily up to maximum tolerated
Period: Overall Study
Arm/Group | Pramipexole | Ropinirole
Started | 121 | 125
Completed | 92 | 97
Not Completed | 29 | 28
Not completed — Adverse Event | 18 | 16
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Other reason (not specified) | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Ropinirole | Total
Number analyzed (Participants) | 121 | 125 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.3) | 59.1 (8.7) | 58.3 (9.0)
Age, Customized [Number; unit: Participants]
  < 50 years | 23 | 17 | 40
  50 to < 65 years | 71 | 74 | 145
  65 to < 75 years | 21 | 30 | 51
  >= 75 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 79 | 78 | 157
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 7 | 3 | 10
  White | 113 | 121 | 234
Height [Mean (Standard Deviation); unit: centimeters] — Measurements collected for 120, 125 participants in Pramipexole, Ropinirole respectively
  centimeters | 171.3 (9.2) | 171.6 (12.4) | 171.5 (10.9)
Weight [Mean (Standard Deviation); unit: kilograms] — Measurements collected for 119, 122 participants in Pramipexole, Ropinirole respectively
  kilograms | 81.32 (17.64) | 82.80 (18.39) | 82.07 (18.00)
Duration of Parkinson's disease diagnosis [Mean (Standard Deviation); unit: years] | 0.97 (1.15) | 1.29 (1.70) | 1.13 (1.46)
Hoehn and Yahr stage [Number; unit: Participants] — This scale is an investigator-completed assessment of the degree of complications arising from Parkinson's disease. The scale ranges from 0 (No signs) to 5 (Bedridden)
  Participants
    Stage 0 | 0 | 0 | 0
    Stage 1 | 28 | 23 | 51
    Stage 1.5 | 11 | 19 | 30
    Stage 2 | 71 | 71 | 142
    Stage 2.5 | 8 | 5 | 13
    Stage 3 | 3 | 7 | 10
    Stage 4 | 0 | 0 | 0
    Stage 5 | 0 | 0 | 0
Alcohol history [Number; unit: Participants]
  Does not drink | 46 | 49 | 95
  Has an average consumption | 75 | 76 | 151
  Fulfills criteria for Abuse/Dependence | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Expert Panel Overall Assessment Following 2 Years on Drug
Description: Expert panel of ophthalmologists assessed retinal deterioration by a review of the components of the comprehensive ophthalmology assessments
Time Frame: up to 2 years
Population: FAS LOCF - full analysis set with last observation carry forward
Measure: Number; unit: Participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 115 | 119
Participants
  Have retinal deterioration | 34 | 33
  Have no retinal deterioration | 81 | 86
Statistical Analysis 1: Comparison: Pramipexole vs Ropinirole; Test type: Superiority or Other; Risk Ratio (RR) = 1.07, 95% CI [0.71 to 1.60]

2. Secondary Outcome: Expert Panel Overall Assessment Following 1 Year on Drug
Description: as for outcome 1
Time Frame: up to 1 years
Population: FAS LOCF - full analysis set with last observation carry forward
Measure: Number; unit: Participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 115 | 119
Participants
  Have retinal deterioration | 28 | 21
  Have no retinal deterioration | 87 | 98

3. Secondary Outcome: Hoehn and Yahr Scale at Baseline
Description: This scale is an investigator-completed assessment of the degree of complications arising from Parkinson's disease. The scale ranges from 0 (No signs) to 5 (Bedridden)
Time Frame: Baseline
Population: TS - treated set
Measure: Number; unit: Participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Participants
  Stage 0 | 0 (0) | 0 (0)
  Stage 1 | 28 | 23
  Stage 1.5 | 11 | 19
  Stage 2 | 71 | 71
  Stage 2.5 | 8 | 5
  Stage 3 | 3 | 7
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

4. Secondary Outcome: Hoehn and Yahr Scale at 1 Year
Description: as for outcome 3
Time Frame: Up to 1 year
Population: TS - treated set
Measure: Number; unit: Participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Participants
  Stage 0 | 1 (1) | 1 (1)
  Stage 1 | 33 | 22
  Stage 1.5 | 9 | 16
  Stage 2 | 70 | 72
  Stage 2.5 | 8 | 8
  Stage 3 | 0 | 6
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

5. Secondary Outcome: Hoehn and Yahr Scale at 2 Years
Description: as for outcome 3
Time Frame: Up to 2 years
Population: TS - treated set
Measure: Number; unit: Participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Participants
  Stage 0 | 1 (1) | 0 (0)
  Stage 1 | 27 | 23
  Stage 1.5 | 6 | 12
  Stage 2 | 74 | 73
  Stage 2.5 | 10 | 10
  Stage 3 | 3 | 7
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

6. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part II, Total Score at Baseline
Description: Part II of the UPDRS collected retrospective information on patient functioning in various activities of daily living. Individual items scored from 0 (Normal) to 4 (Extreme dysfunction). The total score ranged from 0 to 52.
Time Frame: Baseline
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 8.0 (3.8) | 9.5 (4.7)

7. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part II, Total Score at 1 Year
Description: as for outcome 6
Time Frame: 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 7.0 (4.3) | 8.4 (5.0)

8. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part II, Change From Baseline in Total Score at 1 Year
Description: as for outcome 6
Time Frame: Baseline, 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | -1.1 (3.4) | -1.1 (3.6)

9. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part II, Total Score at 2 Years
Description: as for outcome 6
Time Frame: 2 years
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 8.4 (4.6) | 9.3 (5.2)

10. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part II, Change From Baseline in Total Score at 2 Years
Description: as for outcome 6
Time Frame: Baseline, 2 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 0.4 (3.7) | -0.2 (4.0)

11. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part III, Total Score at Baseline
Description: Part III of the UPDRS contained the clinician-scored motor evaluation. Individual items scored from 0 (Normal) to 4 (Extreme dysfunction). The total score ranged from 0 to 56.
Time Frame: Baseline
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 20.7 (9.3) | 22.4 (10.2)

12. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part III, Total Score at 1 Year
Description: as for outcome 11
Time Frame: 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 17.7 (9.3) | 19.8 (10.9)

13. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part III, Change From Baseline in Total Score at 1 Year
Description: as for outcome 11
Time Frame: Baseline, 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | -3.0 (7.2) | -2.6 (6.1)

14. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part III, Total Score at 2 Years
Description: as for outcome 11
Time Frame: 2 years
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 19.7 (9.9) | 20.9 (10.3)

15. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Part III, Change From Baseline in Total Score at 2 Years
Description: as for outcome 11
Time Frame: Baseline, 2 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | -1.0 (7.9) | -1.5 (7.7)

16. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts II and III, Total Score at Baseline
Description: This is the sum of Part II and Part III of the UPDRS. The total score ranged from 0 (Normal) to 108 (Extreme dysfunction).
Time Frame: Baseline
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 28.8 (11.6) | 31.9 (13.4)

17. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts II and III, Total Score at 1 Year
Description: as for outcome 16
Time Frame: 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 24.7 (11.8) | 28.2 (14.5)

18. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts II and III, Change From Baseline in Total Score at 1 Year
Description: as for outcome 16
Time Frame: Baseline, 1 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | -4.1 (8.9) | -3.7 (8.2)

19. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts II and III, Total Score at 2 Years
Description: as for outcome 16
Time Frame: 2 years
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | 28.1 (12.9) | 30.2 (14.1)

20. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS), Parts II and III, Change From Baseline in Total Score at 2 Years
Description: as for outcome 16
Time Frame: Baseline, 2 year
Population: TS - treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 121 | 125
Score on a scale | -0.7 (10.1) | -1.7 (10.5)

21. Secondary Outcome: Clinical Abnormal Findings: Clinical Laboratory Evaluations (Biochemistry and Haematology)and Vital Signs
Description: Clinical relevant abnormalities for clinical laboratory evaluations Biochemistry and Haematology) and Vital Signs. New abnormal findings or worsening of baseline conditions were reported.
Time Frame: Screen (Baseline) and final visit (24 months)
Population: TSlab - treated set with non-missing laboratory evaluations
Measure: Number; unit: participants
Arm/Group | Pramipexole | Ropinirole
Number analyzed (Participants) | 109 | 110
participants
  Haematocrit - Decrease | 1 | 2
  Haemoglobin - Decrease | 8 | 5
  Eosinophils - Increase | 4 | 0
  Phosphate - Decrease | 0 | 2
  Calcium - Increase | 1 | 0
  Glucose - Decrease | 4 | 0

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | Pramipexole | Ropinirole
Serious Adverse Events (participants affected / at risk) | 22/121 | 21/125
Other Adverse Events (participants affected / at risk) | 97/121 | 101/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=121) | Ropinirole (N=125)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain mass (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Hyperthecosis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=121) | Ropinirole (N=125)
Vision blurred (Eye disorders) | 7 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 18 | 26
Diarrhoea (Gastrointestinal disorders) | 6 | 9
Dry mouth (Gastrointestinal disorders) | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 8
Nausea (Gastrointestinal disorders) | 31 | 59
Vomiting (Gastrointestinal disorders) | 3 | 12
Chest pain (General disorders) | 6 | 7
Fatigue (General disorders) | 27 | 25
Oedema peripheral (General disorders) | 22 | 18
Nasopharyngitis (Infections and infestations) | 17 | 16
Sinusitis (Infections and infestations) | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 12 | 13
Urinary tract infection (Infections and infestations) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 13
Dizziness (Nervous system disorders) | 27 | 35
Dizziness postural (Nervous system disorders) | 9 | 9
Headache (Nervous system disorders) | 15 | 27
Hypoaesthesia (Nervous system disorders) | 5 | 9
Paraesthesia (Nervous system disorders) | 0 | 10
Somnolence (Nervous system disorders) | 53 | 71
Sudden onset of sleep (Nervous system disorders) | 11 | 16
Abnormal dreams (Psychiatric disorders) | 8 | 7
Anxiety (Psychiatric disorders) | 10 | 14
Depression (Psychiatric disorders) | 8 | 15
Insomnia (Psychiatric disorders) | 19 | 27
Sleep disorder (Psychiatric disorders) | 9 | 10
Erectile dysfunction (Reproductive system and breast disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 6 | 10
Hypertension (Vascular disorders) | 9 | 10
Orthostatic hypotension (Vascular disorders) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.